CLINICAL TRIAL: NCT03409627
Title: A Phase I, Open Label, Safety Study of INXN-4001 Delivered Via Retrograde Coronary Sinus Infusion in Patients With an Outpatient Left Ventricular Assist Device (LVAD)
Brief Title: Novel INXN-4001 Triple Effector Plasmid in Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Triple-Gene, LLC (Industry)
Collaborators: Intrexon Corporation (Industry); Precigen, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INXN-4001-001
Record Dates: First submitted 2017-11-03; First posted 2018-01-24 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure; Cardiovascular Diseases; Heart-Assist Device
Keywords: retrograde coronary sinus infusion; DNA; non-viral; triple effector plasmid; gene therapy; regenerative medicine; non-stem cell
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Single infusion of INXN-4001, Dose 1
  Interventions: Biological: INXN-4001
- Group 2 (Experimental): Single infusion of INXN-4001, Dose 2
  Interventions: Biological: INXN-4001

INTERVENTIONS:
Biological: INXN-4001 — Retrograde coronary sinus infusion of triple effector plasmid (INXN-4001)

SUMMARY:
To evaluate the safety of retrograde coronary sinus infusion (RCSI) of a novel triple-effector plasmid (INXN-4001) in outpatient LVAD recipients as assessed by incidence of all study intervention-related adverse events occurring up to 6 months post-RCSI (primary endpoints), and to evaluate general safety by assessing incidence of cardiac specific adverse events and the incidence of related serious adverse events at intervals up to 12 months post-infusion (or until cardiac transplantation or death).

DETAILED DESCRIPTION:
This is a first-in-human, phase I, open label, safety study of INXN-4001 delivered via RCSI in patients with outpatient LVAD. Twelve stable patients with implanted LVAD for mechanical support of end stage heart failure have been allocated into 2 cohorts (6 subjects each) to evaluate the safety of infusing the same amount of INXN-4001 (80mg) in 2 volumes (40mL and 80mL) at 20mL/min rate. Ongoing safety assessments include clinical labs, physical exams, ECG and medical history collected during clinic visits at: pre-treatment, day 3, then 1, 3, 6, 9, and 12 months after dosing via RCSI. During visits, subjects complete the KCCQ questionnaire and are evaluated via 6-min walk test (6MWT) prior to and during an LVAD wean interval. Daily activity data is collected throughout the study using a wearable biosensor (Actigraph).

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients with a stable LVAD implanted for end-stage heart failure
* Must be managed in an outpatient setting and on stable medication regimen

Exclusion Criteria:

* Women who are pregnant or nursing
* Patients who have been on another clinical trial for heart failure in the last 90 days, or have received any stem cell or gene therapy within the previous year.
* Patient is not able to complete a Six Minute Walk Test or unable to tolerate an LVAD wean in the past 3 months
* Patient has an active infection requiring systemic antibiotics or an autoimmune disease requiring systemic immunosuppressants
* Patient has a history of arrhythmia, uncontrolled diabetes, diabetic retinopathy, systemic lupus erythematosus, macular degeneration, hyper-coagulation, or stroke
* Patient has had a myocardial infarction related to ischemia within the past 30 days
* Patient has had certain prior surgeries such as organ transplant, cardiac transplantation, left ventricle reduction surgery, or cardiomyoplasty
* Patient has infectious disease, such as hepatitis B or C, or human immunodeficiency virus (HIV)
* Patient has a history of cancer within the past 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and feasibility of INXN-4001 | 6 months
  As assessed by incidence of all study intervention-related adverse events occurring up to 6 months post- treatment intervention-related adverse events

SECONDARY OUTCOMES:
Wean tolerability following treatment with INXN-4001 | 12 months
  Improvement in 6 minute walk duration and distance
Quality of Life following treatment with INXN-4001 | 12 months
  Change in Kansas City Cardiomyopathy Questionnaire responses
Feasibility of biosensor activity tracking | 12 months
  Ability to collect daily activity level as measured by wearable biosensor
Overall safety of INXN-4001 | 12 months
  Incidence of cardiac-specific adverse events and study intervention-related serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: David Bull, MD, Principal Investigator — University of Arizona; Ulrich Jorde, MD, Principal Investigator — Montefiore Medical Center; Gregory Egnaczyk, MD, Principal Investigator — The Christ Hospital
Locations (2):
- United States (2):
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - The Lindner Research Center, The Christ Hospital Health Network, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No